CLINICAL TRIAL: NCT00239772
Title: Cognitive Processes in PTSD: Treatment
Brief Title: Cognitive Processing Therapy Versus Prolonged Exposure for Treating Women With Post-Traumatic Stress Disorder Brought on by Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, St. Louis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH051509-05 (NIH); R01MH051509-05 (NIH); DSIR AT-AS
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Cognitive Therapy; PTSD; Females; Rape; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy
Behavioral: Prolonged Exposure Therapy

SUMMARY:
This study will evaluate the effectiveness of cognitive processing therapy versus prolonged exposure therapy in treating women with post-traumatic stress disorder (PTSD) brought on by sexual assault.

DETAILED DESCRIPTION:
PTSD is a psychiatric disorder that can occur following exposure to a traumatic event in which grave physical harm occurred or was threatened. PTSD is marked by clear biological changes as well as psychological symptoms. Many people with PTSD repeatedly relive the trauma in the form of flashback episodes, memories, nightmares, or frightening thoughts. This study will evaluate the effectiveness of cognitive processing therapy (CPT) versus prolonged exposure therapy in treating women with PTSD brought on by sexual assault.

Participants in this single-blind study will be randomly assigned to one of three conditions: CPT, prolonged exposure therapy (PE), or minimal attention (MA). Individuals assigned to receive CPT will attend therapy sessions twice weekly for 6 weeks. Each session will be 1 hour long, except for sessions 4 and 5, which will be 1.5 hours long. CPT will focus on helping each individual to process accurate memories of the traumatic event and to work through any memories that cannot be completely ignored, nor completely integrated back into their thinking. Also included in CPT will be an exposure component, in which participants will be encouraged to recall the traumatic event and experience any emotions connected to it. Participants assigned to receive PE therapy will attend an initial 1-hour therapy session, followed by 4 weeks of additional sessions that will meet twice weekly. Each of these 8 sessions will be 1.5 hours long. PE will entail oral exposure without modification of the participant's cognitions. Participants will discuss their traumatic experiences in detail during each session to aid in emotional processing. All PE sessions will be audio taped. Participants will listen to the tapes of their sessions on their own to further assist with emotional processing. Individuals assigned to receive MA will receive no therapy for the first 6 weeks. At the end of this initial phase, they will be assigned to receive either CPT or PE if they still meet diagnostic criteria for PTSD. Symptoms of PTSD, feelings of guilt and shame, and overall perception of self and surroundings will be assessed at baseline, post-treatment, and at follow-up visits at 3, 6, and 9 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one incidence of rape
* Diagnosed with post-traumatic stress disorder

Exclusion Criteria:

* Rape occurred before the age of 13 and was committed by a family member
* Rape was committed by a spouse who is currently living in the same household
* Psychosis
* Mental retardation
* Current pathology that may complicate symptoms of post-traumatic stress disorder
* Currently suicidal or parasuicidal
* Currently addicted to drugs or alcohol
* Illiterate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1994-05

PRIMARY OUTCOMES:
Post-traumatic stress disorder symptoms; measured immediately post-treatment and at 3, 6, and 9 months post-treatment

SECONDARY OUTCOMES:
Feelings of guilt and shame; measured immediately post-treatment and at 3, 6, and 9 months post-treatment
Overall perception of self and surroundings; measured immediately post-treatment and at 3, 6, and 9 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Resick, PhD, Principal Investigator — National Center for PTSD, Women's Health Sciences Division
Locations (1):
- Center for Trauma and Recovery, University of Missouri - St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270